CLINICAL TRIAL: NCT02315235
Title: The Efficacy and Safety of Peripheral Mobilized Mononuclear Cell-based Therapy in Patients With Diabetic Painful Neuropathy
Brief Title: The Peripheral Mobilized Mononuclear Cell-based Therapy in Patient With Diabetic Neuropathy
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Do not have a sutable subjects.
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Hye Seung Jung, Associate professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: mononuclear cell-based therapy
Record Dates: First submitted 2014-12-05; First posted 2014-12-11 (Estimated); Last update posted 2016-04-15 (Estimated); Status verified 2016-04

CONDITIONS: Diabetic Neuropathy
MeSH Terms: conditions — Diabetic Neuropathies | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- control (Active Comparator): The operator inject normal saline(control) to thirty site of the other side leg of active comparator. The volume of one site injection is 0.5 ml. The depth of needle injection would be 1.5cm.
  Interventions: Biological: Normal saline
- stem cell (mononuclear cell) (Active Comparator): The stem cell (mononuclear cell) is injected to thirty site of one side leg in operating room after general anesthesia. The volume of one site injection is 0.5 to 1.0 ml. The depth of needle injection would be 1.5cm.
  Interventions: Biological: stem-cell

INTERVENTIONS:
Biological: Normal saline — Normal saline is injected in one leg of patient.
  Arms: control
Biological: stem-cell — Granulocyte colony-stimulating factor (G-CSF) is injected into subcutaneous for three days prior to the blood collection (D-3 to D-1). Peripheral mononuclear stem-cell is collected by Cobe spectra apheresis system in D-day.
  The stem-cell (mononuclear cell) is injected into the muscle in the other side leg of patient.
  Arms: stem cell (mononuclear cell)

SUMMARY:
To investigate the efficacy and safety of autologous peripheral blood stem cell based therapy in patients with diabetic painful neuropathy.

DETAILED DESCRIPTION:
Diabetic painful neuropathy a prevalent, disabling disorder. Currently, the only effective treatments are glucose control and pain management. Diabetic neuropathy is characterized by reduction of vascularity in peripheral nerves and deficiency in neurotrophic and angiogenic factors. Recent studies have shown that bone marrow (BM)-derived stem or progenitor cells have favorable effects on the repair of cardiovascular diseases. Since these BM-derived stem or progenitor cells contain various angiogenic and neurotrophic factors, these cells have been attempted for treating experimental diabetic neuropathy, and turned out to be effective for reversing various manifestations of experimental diabetic neuropathy.

However, stem-cell therapy was not proven in human study. Therefore, we will investigate the efficacy and safety of autologous peripheral blood stem cell injection in diabetic neuropathy.

ELIGIBILITY:
Inclusion Criteria:

* symptomatic diabetic neuropathy moderate pain more than 3 months Michigan Neuropathy Screening Instrument (MNSI) >3 3/day mean pain scale > NRS 4 Body weight >50 kg systolic blood pressure: 90-150 mmHg, Diastolic blood pressure <100 mmHg, Body temperature <37.5℃, Pulse rate: 50-100/min

Exclusion Criteria:

* other cause of neuropathy symptomatic peripheral vessel disease skin lesion or arthritis central neuronal disease drug addiction or abuse Aspartate aminotransferase or Alanine aminotransferase >1.5 times than upper normal limit range Creatinine clearance rate <60ml/min or dialysis Myocardial infarction, unstable angina or heart failure diagnosed in 3 months psychologic disorder pregnancy or lactation

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-05; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Estimated)

PRIMARY OUTCOMES:
Changes in pain for a week after the procedure | baseline, 4 week, 12 week
  The pain scale was calculate by Numeric rating scale (NRS). We observe a change in NRS pain scores during the follow-up period.

SECONDARY OUTCOMES:
The evaluation of changes in the specific neuro-sensory system | baseline, 4 week, 12 week
  The following tests was evaluated during the follow-up period. The pain intensity was evaluated by short-form McGill Pain Questionnaire and by sleep disturbance pain score. The quantitative change of sensory nerve was evaluated by quantitative sensory test (QST). We measure serum neuron-specific enolase (NSE), glucose, insulin and c-peptide. The amount of drug requirements will also assess at each follow-up period.

OTHER OUTCOMES:
The secondary effect of the procedure for the peripheral nerves and blood vessels | baseline, 12 week
  Michigan neuropathy screening instrument (MNSI) is used for screening for diabetic peripheral neuropathy. Changes in patient's mood is assessed by the Beck Depression Inventory (BDI) system. Electrophysiological tests are used in the evaluation of nerve conduct velocity. Skin punch biopsy is used to evaluate the density of epidermal nerve fibers. Improvement of blood flow in the peripheral veins is evaluated by ankle brachial index (ABI), pulse wave velocity (PWV) and digital arterial plethysmography. We measure serum glucose, insulin ant c-peptide. The amount of drug requirements will also assess at each follow-up period.

CONTACTS AND LOCATIONS:
Overall Officials: Hye Seung Jung, Ph.D., Study Chair — Seoul Nation University Hospital
Locations (1):
- SeoulNUH, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No